CLINICAL TRIAL: NCT02307084
Title: An Investigation Into the Efficacy of Pre-operative Long Saphenous Vein Mapping Using Ultrasound for Use in Coronary Artery Bypass Grafting to Reduce Vein Harvest Site Complications.
Brief Title: Ultrasound to Prevent Leg Wound Complications in Heart Bypass.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of Chief Investigator/Principal Investigator
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CS/2014/4661
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Surgical Wound Infection; Coronary Artery Bypass
Keywords: surgical site infection; long saphenous vein; coronary artery bypass grafting
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-operative ultrasound imaging (Experimental): Subjects that are randomly allocated to this group will have ultrasound imaging assessment of the long saphenous vein in both legs. This will allow assessment of the suitability of the long saphenous vein and marking of the distribution prior to heart bypass surgery to allow targeted harvesting of a bypass conduit.
  Interventions: Procedure: Ultrasound imaging of the long saphenous vein
- Current protocol (No Intervention): This group will not undergo pre-operative ultrasound imaging of the long saphenous vein in accordance with current Trust protocols.

INTERVENTIONS:
Procedure: Ultrasound imaging of the long saphenous vein — Ultrasound imaging of the long saphenous vein from the ankle to the saphenofemoral junction. This will allow assessment of vein calibre, branches and bifurcations, presence of thrombophlebitis and distribution. The presence of a proximal deep vein thrombosis will also be assessed.
  Arms: Pre-operative ultrasound imaging

SUMMARY:
The long saphenous vein is traditionally harvested for use as a conduit in coronary artery bypass grafting surgery. Currently, the long saphenous vein is not imaged prior to surgery. This study aims to evaluate preoperative ultrasound mapping of the long saphenous vein to to improve patient and clinical outcomes.

DETAILED DESCRIPTION:
A vein from the leg is widely is widely harvested during coronary artery bypass grafting (CABG) surgery for bypass of diseased coronary arteries. This vein is called the long saphenous vein.

Currently, the long saphenous vein (LSV) is harvested blind by surgical practitioners with no imaging prior to surgery to decide on whether this vein is suitable for use in heart bypass surgery. This can result in fruitless incisions and result in additional unnecessary surgical wounds in the leg(s) to identify a suitable section of vein that can be used in the bypass operation. In these cases, excessive surgical trauma to the leg can increase the risk of a wound infection.

There is some evidence that ultrasound imaging of the LSV improves leg wound outcomes in patients having CABG surgery. Some studies have reported reductions in vein wound infection rates, vein harvest time, length of hospitalisation and length of wounds.

The purpose of this study will be to investigate the potential benefit of ultrasound imaging as a randomised control trial. One group will have ultrasound imaging of the long saphenous vein prior to heart bypass surgery. A second group will not undergo ultrasound imaging which is current practice at the Bristol Heart Institute.

Ultrasound imaging of the long saphenous vein will allow planning and selection of the most optimal segment of vein. This targeted approach will allow guidance of surgical incisions away from unsuitable segments and thus potentially improving leg wound outcomes.

The primary endpoint for this study will be to assess leg wound infection between the two randomised groups. Other endpoints that will be assessed are patient satisfaction, wound length, time taken to remove the vein, blood loss from the leg wound during surgery and the number of wounds in your leg.

ELIGIBILITY:
Inclusion Criteria:

* Listed for CABG surgery with long saphenous vein harvesting.
* Aged over 18 years.
* Capable of providing informed consent.
* Five days or more to consider participation prior to surgery if an outpatient or 2 days if an inpatient referred by their consultant.
* Operative procedure to be undertaken at the Bristol Heart Institute.

Exclusion Criteria:

* Operation within 48h hours if an inpatient or 5 days if an outpatient.
* Aged below 18 years of age.
* Incapable of providing informed consent i.e. confirmed diagnosis of dementia or other mental health conditions or unconscious.
* Current participant in a different randomised control trial.
* Pregnancy
* Active cancer
* Immunosuppressed.
* Non-English speaker that requires a Trust translator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Surgical site infection at the conduit harvest site | 30 days of CABG surgery
  The ASEPSIS tool is a well established tool to quantify wound healing disturbances.

SECONDARY OUTCOMES:
Ability to identify abnormal segments of vein on ultrasound and direct surgical excision away from such areas. | baseline
  Applicable to the ultrasound imaged group only. The incidence of an abnormal segment of vein will be quantified and whether or not this has led to avoidance of unnecessary surgical excisions.
Time taken to harvest a suitable conduit. | intraoperative
  The time to harvest a suitable conduit will be recorded during CABG surgery.
Length of lower limb vein harvest wounds. | 1 day Post-operation
  Length of conduit harvest wounds will be measured after surgery to the nearest centimetre.
Blood loss from the vein harvest wound | intraoperative
  The blood loss from the conduit harvest wound(s) will be measured during surgery by weighing swabs.
Patient questionnaire to assess wound/scar satisfaction and complications. | 30 days from surgery
  An assessment of patient satisfaction and non-infective complications related to the conduit harvesting for CABG surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Reshat Reshat, PhD, Principal Investigator — University Hospital Bristol NHS FT; Teresa Robinson, MSc, Study Director — University Hospital Bristol NHS FT
Locations (1):
- University Hospital Bristol NHS FT, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No